CLINICAL TRIAL: NCT00076999
Title: Multiple-dose, Open-label, Randomized, Safety and Pharmacokinetic Study of Tipranavir in Combination With Low-dose Ritonavir in HIV-infected Pediatric Patients
Brief Title: Pharmacokinetics and Safety Study of Tipranavir in Combination With Low Dose Ritonavir in Human Immunodeficiency Virus (HIV)-Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.14
Record Dates: First submitted 2004-02-09; First posted 2004-02-10 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir

ARMS (2):
- TPV/r 290/115 mg/m^2 (Experimental): TPV and RTV oral solution low dose
  Interventions: Drug: TPV oral solution; Drug: RTV oral solution
- TPV/r 375/150 mg/m^2 (Experimental): TPV and RTV oral solution high dose
  Interventions: Drug: TPV oral solution; Drug: RTV oral solution

INTERVENTIONS:
Drug: TPV oral solution — Tipranavir oral solution
  Arms: TPV/r 290/115 mg/m^2
Drug: TPV oral solution — Tipranavir oral solution
  Arms: TPV/r 375/150 mg/m^2
Drug: RTV oral solution — Ritonavir oral solution
  Arms: TPV/r 290/115 mg/m^2
Drug: RTV oral solution — Ritonavir oral solution
  Arms: TPV/r 375/150 mg/m^2

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of tipranavir (TPV) oral formulation and soft gelatin capsules together with low-dose ritonavir in HIV-infected children and adolescents, to provide information concerning the pharmacokinetic characteristics of tipranavir and ritonavir in this age group, and to determine the relative bioavailability of the TPV liquid formulation and TPV capsule formulation in adolescents switching from liquid to capsule.

The secondary objective of this study is the determination of the dose of topranavir and ritonavir (TPV/r) in children and adolescents between 2 and 18 years of age required for an adult equivalent systemic exposure of TPV/r 500 mg / 200 mg.

ELIGIBILITY:
Inclusion criteria:

1. Males and females between 2 and 18 years of age.
2. A confirmed diagnosis of HIV-1 infection as defined by two positive assays from two different samples taken at least two weeks apart. The two results may be any combination of the following:

   HIV ribonucleic acid (RNA) detected by reverse transcriptase (RT)-polymerase chain reaction(PCR) or HIV proviral deoxyribonucleic acid (DNA) detected by PCR HIV culture p24 antigen detection Licensed HIV enzyme-linked immunosorbent assay (ELISA) with confirmatory Western blot
3. Viral load > 1500 RNA copies/mL.
4. Acceptable screening laboratory values indicative of adequate baseline organ function. Laboratory values are considered acceptable if severity is no higher than Grade 1 for all tests defined by the Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading Severity of Pediatric Adverse Experiences (> 3 months of age) with the following exceptions:

   Grade 2 gamma-glutamyl transferase Grade 2 cholesterol Grade 2 triglycerides
5. Signed informed consent prior to study participation from the patient or a legal guardian.

   Active assent must be given by the patient if the child and/or adolescent is capable of understanding the provided study information (this applies to children with the intellectual age of 7 years or greater)
6. In the opinion of the investigator, an ability to take medications and comply with the requirements of the protocol.

Exclusion criteria:

1. Female patients of childbearing potential who:

   have a positive serum pregnancy test at screening are breast feeding are planning on becoming pregnant are not willing to use two methods of contraception to include at least one barrier method (e.g. latex condom plus spermicidal jelly/foam)
2. Active hepatitis B or C disease defined as hepatitis B surface antigen (HBsAg) positivity or hepatitis C (HCV) antibody or RNA positivity with aspartate aminotransferase(AST)/ alanine aminotransferase(ALT) > Grade 2.
3. Life expectancy < 12 months.
4. Patients who are unwilling to abstain from ingesting contraindicated medications and substances which may significantly affect plasma levels of the study medications, notably:

   Grapefruit juice or Seville oranges Herbal preparations containing St. John's Wort or milk thistle Garlic supplements
5. Active substance abuse.
6. Use of investigational medications or vaccines within 28 days before study entry or during the trial. Some expanded access antiretroviral medications may be acceptable, but must be approved by sponsor.
7. Requirement for any therapy for malignancy or immunomodulatory drug (e.g. interferon, cyclosporine, hydroxyurea, interleukin-2) within 28 days of study entry. Replacement intravenous gamma globulin treatment is acceptable.
8. Any active opportunistic infection within 28 days before study entry or other clinically significant findings that may compromise the outcome of the study.
9. Patients with malabsorption, severe chronic diarrhea or vomiting (more than two episodes of moderate or severe intensity, not attributed to medication therapy and lasting more than four days) within 28 days of the study.
10. Evidence or symptoms of encephalopathy or developmental delay that would reduce compliance.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2003-11; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (30):
- United States (9):
  - 1182.14.00001 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1182.14.00006 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1182.14.00010 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 1182.14.00004 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1182.14.00008 Boehringer Ingelheim Investigational Site, North Worcester, Massachusetts
  - 1182.14.00009 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1182.14.00002 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 1182.14.00007 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1182.14.00003 Boehringer Ingelheim Investigational Site, Houston, Texas
- 1182.14.5401 Fundación Huésped, Capital Federal, Argentina
- Brazil (2):
  - 1182.14.55002, São Paulo
  - 1182.14.55003, São Paulo
- Canada (2):
  - 1182.14.11002 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1182.14.11001 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- France (6):
  - 1182.14.33004 Boehringer Ingelheim Investigational Site, Lyon
  - 1182.14.33005 Boehringer Ingelheim Investigational Site, Nantes
  - 1182.14.33001 Boehringer Ingelheim Investigational Site, Paris
  - 1182.14.33002 Boehringer Ingelheim Investigational Site, Paris
  - 1182.14.33003 Boehringer Ingelheim Investigational Site, Paris
  - 1182.14.33006 Boehringer Ingelheim Investigational Site, Paris
- Germany (3):
  - 1182.14.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1182.14.49001 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1182.14.49004 Boehringer Ingelheim Investigational Site, München
- Italy (2):
  - 1182.14.39001 Boehringer Ingelheim Investigational Site, Padua
  - 1182.14.39003 Boehringer Ingelheim Investigational Site, Roma
- Mexico (2):
  - 1182.14.52001 CLINDI (Clínica de Inmunodeficiencias), México, D.F.
  - 1182.14.52002, México, D.F.
- 1182.14.00005 Boehringer Ingelheim Investigational Site, San Juan, Puerto Rico
- Spain (2):
  - 1182.14.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.14.34001 Boehringer Ingelheim Investigational Site, Madrid

REFERENCES:
- [Derived] Salazar JC, Cahn P, Della Negra M, De Aquino MZ, Robinson PA, Jelaska A, Mikl J. Efficacy and safety of tipranavir coadministered with ritonavir in HIV-1-infected children and adolescents: 5 years of experience. Pediatr Infect Dis J. 2014 Apr;33(4):396-400. doi: 10.1097/INF.0000000000000038. PMID 23995585
- [Derived] Salazar JC, Cahn P, Yogev R, Negra MD, Castelli-Gattinara G, Fortuny C, Flynn PM, Giaquinto C, Ruan PK, Smith ME, Mikl J, Jelaska A; PACTG 1051/BI Study Team. Efficacy, safety and tolerability of tipranavir coadministered with ritonavir in HIV-1-infected children and adolescents. AIDS. 2008 Sep 12;22(14):1789-98. doi: 10.1097/QAD.0b013e32830c481b. PMID 18753862

RESULTS

PARTICIPANT FLOW:
Groups:
- TPV OS 2-<6 Yrs: Tipranavir Oral Solution (TPV OS), ages 2-5
- TPV OS 6-<12 Yrs: Tipranavir Oral Solution (TPV OS), ages 6-11
- TPV OS 12-18 Yrs: Tipranavir Oral Solution (TPV OS), ages 12-18
- TPV SEDDS 6-<12 Yrs: TPV self-emulsifying drug delivery system (SEDDS), ages 6-11
- TPV SEDDS 12-18 Yrs: TPV self-emulsifying drug delivery system (SEDDS), ages 12-18
Period: Overall Study
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 6-<12 Yrs | TPV SEDDS 12-18 Yrs
Started | 25 | 31 | 19 | 6 | 34
Completed | 13 | 7 | 2 | 5 | 9
Not Completed | 12 | 24 | 17 | 1 | 25
Not completed — Adverse Event | 2 | 8 | 6 | 0 | 2
Not completed — Protocol Violation | 0 | 3 | 4 | 0 | 9
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 3 | 0 | 1
Not completed — Other reason (not specified) | 8 | 8 | 4 | 1 | 13

BASELINE CHARACTERISTICS:
Groups:
- TPV OS 2-<6 Yrs: Patients treated with Tipranavir Oral Solution, ages 2-5
- TPV OS 6-<12 Yrs: Patients treated with Tipranavir Oral Solution, ages 6-11
- TPV OS 12-18 Yrs: Patients treated with Tipranavir Oral Solution, ages 12-18
- TPV SEDDS 12-18 Yrs: Patients treated with Tipranavir SEDDS, ages 12-18
- Total: Total of all reporting groups
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs | Total
Number analyzed (Participants) | 25 | 37 | 24 | 29 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.1 (1.1) | 9.5 (1.4) | 14.4 (1.7) | 15.1 (1.7) | 10.8 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 10 | 15 | 50
  Male | 15 | 22 | 14 | 14 | 65
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic / Latino | 22 | 20 | 11 | 8 | 61
  Mixed Race | 1 | 0 | 2 | 2 | 5
  Unknown | 2 | 17 | 11 | 19 | 49
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18 | 26 | 16 | 20 | 80
  Black | 6 | 10 | 8 | 9 | 33
  Asian | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  North America | 3 | 14 | 13 | 11 | 41
  South America and Mexico | 22 | 14 | 4 | 5 | 45
  Europe | 0 | 9 | 7 | 13 | 29
Antiretroviral Experienced [Number; unit: participants]
  Yes | 24 | 36 | 24 | 28 | 112
  No | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Number Patients With at Least 1 log10 Viral Load Reduction From Baseline at Week 24 (Non-completers Considered Failures)
Time Frame: baseline, week 24
Population: Full Analysis Set included all patients treated with study medication having at least one on-treatment efficacy assessment
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
participants
  Viral load reduction | 20 | 18 | 9 | 13
  No viral load reduction | 5 | 19 | 15 | 16
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.02, Fisher Exact
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.78, Fisher Exact

2. Secondary Outcome: Number Patients With at Least 1 log10 Viral Load Reduction From Baseline at Week 48 (Non-completers Considered Failures)
Time Frame: baseline, week 48
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
participants
  Viral load reduction | 19 | 14 | 8 | 9
  No viral load reduction | 6 | 23 | 16 | 20
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.00, Fisher Exact
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 1.00, Fisher Exact

3. Secondary Outcome: Number Patients With at Least 1 log10 Viral Load Reduction From Baseline at Week 100 (Non-completers Considered Failures)
Time Frame: baseline, week 100
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
participants
  Viral load reduction | 14 | 13 | 6 | 7
  No viral load reduction | 11 | 24 | 18 | 22
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.12, Fisher Exact
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 1.00, Fisher Exact

4. Secondary Outcome: Number Patients With HIV RNA <400 Copies/mL at Week 24 (Non-completers Considered Failures)
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
participants
  Viral load reduction | 16 | 15 | 8 | 10
  No viral load reduction | 9 | 22 | 16 | 19
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.12, Fisher Exact
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 1.00, Fisher Exact

5. Secondary Outcome: Number Patients With HIV RNA <400 Copies/mL at Week 48 (Non-completers Considered Failures)
Time Frame: baseline, week 48
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
participants
  Viral load reduction | 18 | 13 | 8 | 9
  No viral load reduction | 7 | 24 | 16 | 20
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.01, Fisher Exact
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 1.00, Fisher Exact

6. Secondary Outcome: Number Patients With HIV RNA <400 Copies/mL at Week 100 (Non-completers Considered Failures)
Time Frame: baseline, week 100
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
participants
  Viral load reduction | 14 | 11 | 6 | 7
  No viral load reduction | 11 | 26 | 18 | 22
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.06, Fisher Exact
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 1.00, Fisher Exact

7. Secondary Outcome: Number Patients With HIV RNA <50 Copies/mL at Week 24 (Non-completers Considered Failures)
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
participants
  Viral load reduction | 10 | 12 | 6 | 8
  No viral load reduction | 15 | 25 | 18 | 21
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.60, Fisher Exact
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 1.00, Fisher Exact

8. Secondary Outcome: Number Patients With HIV RNA <50 Copies/mL at Week 48 (Non-completers Considered Failures)
Time Frame: baseline, week 48
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
participants
  Viral load reduction | 13 | 13 | 6 | 8
  No viral load reduction | 12 | 24 | 18 | 21
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.20, Fisher Exact
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 1.00, Fisher Exact

9. Secondary Outcome: Number Patients With HIV RNA <50 Copies/mL at Week 100 (Non-completers Considered Failures)
Time Frame: baseline, week 100
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
participants
  Viral load reduction | 12 | 11 | 5 | 6
  No viral load reduction | 13 | 26 | 19 | 23
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.18, Fisher Exact
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 1.00, Fisher Exact

10. Secondary Outcome: Baseline Median Viral Load log10 Copies/mL
Time Frame: baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
log10 copies/mL | 5.0 (4.5, 5.3) [4.5 to 5.3] | 4.6 (4.4, 5.1) [4.4 to 5.1] | 5.1 (4.0, 5.5) [4.0 to 5.5] | 4.6 [4.1 to 5.0]

11. Secondary Outcome: Median Change From Baseline in Viral Load log10 Copies/mL at Week 24 (Last Observation Carried Forward)
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
log10 copies/mL | -2.5 (-3.0, -1.8) [-3.0 to -1.8] | -1.7 (-2.7. -0.4) [-2.7 to -0.4] | -0.4 (-1.7, 0.0) [-1.7 to 0.0] | -1.1 [-2.3 to 0.0]
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.02, ANOVA
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.47, ANOVA

12. Secondary Outcome: Median Change From Baseline in Viral Load log10 Copies/mL at Week 48 (Last Observation Carried Forward)
Time Frame: baseline, week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
log10 copies/mL | -2.7 (-3.3, -1.5) [-3.3 to -1.5] | -1.0 (-2.4, -0.1) [-2.4 to -0.1] | -0.4 (-1.6, 0.0) [-1.6 to 0.0] | -0.8 [-2.2 to 0.2]
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.00, ANOVA
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.81, ANOVA

13. Secondary Outcome: Median Change From Baseline in Viral Load log10 Copies/mL at Week 100 (Last Observation Carried Forward)
Time Frame: baseline, week 100
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 37 | 24 | 29
log10 copies/mL | -2.7 (-3.3, -1.0) [-3.3 to -1.0] | -1.2 (-2.4, -0.1) [-2.4 to -0.1] | -0.2 (-1.5, 0.0) [-1.5 to 0.0] | -0.4 [-1.9 to 0.2]
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.00, ANOVA
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.69, ANOVA

14. Secondary Outcome: Baseline Median CD4+ Cell Count (Cells/mm3)
Time Frame: baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 23 | 35 | 23 | 29
cells/mm3 | 795 (536,1229) [536 to 1229] | 398 (232,734) [232 to 734] | 208 (100,475) [100 to 475] | 330 [180 to 389]

15. Secondary Outcome: Median Change From Baseline in CD4+ Cell Count (Cells/mm3) at Week 24 (Last Observation Carried Forward)
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 23 | 35 | 23 | 29
cells/mm3 | 293 (27,396) [27 to 396] | 133 (5,217) [5 to 215] | 24 (0, 56) [0 to 56] | 56 [0 to 168]
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.64, ANOVA
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.26, ANOVA

16. Secondary Outcome: Median Change From Baseline in CD4+ Cell Count (Cells/mm3) at Week 48 (Last Observation Carried Forward)
Time Frame: baseline, week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 23 | 35 | 23 | 29
cells/mm3 | 323 (-110,529) [-110 to 529] | 143 (-6,249) [-6 to 249] | 21 (0, 95) [0 to 95] | 39 [-61 to 153]
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.25, ANOVA
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.70, ANOVA

17. Secondary Outcome: Median Change From Baseline in CD4+ Cell Count (Cells/mm3) at Week 100 (Last Observation Carried Forward)
Time Frame: baseline, week 100
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 23 | 35 | 23 | 29
cells/mm3 | 294 (-125,416) [-125 to 416] | 121 (-9,319) [-8 to 319] | 12 (-1,100) [-1 to 100] | 45 [0 to 124]
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.73, ANOVA
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.79, ANOVA

18. Secondary Outcome: Median Baseline CD4 Percent
Description: Percentage of lymphocytes that are CD4 cells
Time Frame: baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 23 | 35 | 23 | 29
percentage of cells | 26 (19, 35) [19 to 35] | 19 (10, 29) [10 to 29] | 12 (8, 21) [8 to 21] | 19 [14 to 25]

19. Secondary Outcome: Median Change From Baseline in CD4 Percent at Week 24 (Last Observation Carried Forward)
Description: Percentage of lymphocytes that are CD4 cells
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 23 | 35 | 23 | 29
percentage of cells | 7 (2, 10) [2 to 10] | 4 (0.8) [0 to 8] | 1 (0.4) [0 to 4] | 2 [0 to 6]
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.38, ANOVA
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.20, ANOVA

20. Secondary Outcome: Median Change From Baseline in CD4 Percent at Week 48 (Last Observation Carried Forward)
Description: Percentage of lymphocytes that are CD4 cells
Time Frame: baseline, week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 23 | 35 | 23 | 29
percentage of cells | 7 (2, 13) [2 to 13] | 5 (0.8) [0 to 8] | 1 (0.5) [0 to 5] | 3 [-1 to 6]
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.08, ANOVA
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.36, ANOVA

21. Secondary Outcome: Median Change From Baseline in CD4 Percent at Week 100 (Last Observation Carried Forward)
Description: Percentage of lymphocytes that are CD4 cells
Time Frame: baseline, week 100
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 23 | 35 | 23 | 29
percentage of cells | 6 (3, 10) [3 to 10] | 4 (0.9) [0 to 9] | 1 (0.7) [0 to 7] | 0 [-2 to 7]
Statistical Analysis 1: Comparison: TPV OS 2-<6 Yrs vs TPV OS 6-<12 Yrs; Comparison of TPV OS 2-<6 yrs versus TPV OS 6-<12 yrs; Test type: Superiority or Other; p = 0.23, ANOVA
Statistical Analysis 2: Comparison: TPV OS 12-18 Yrs vs TPV SEDDS 12-18 Yrs; Comparison of TPV OS 12-18 yrs versus TPV SEDDS 12-18 yrs; Test type: Superiority or Other; p = 0.23, ANOVA

22. Secondary Outcome: Number Patients With Compliance With Tipranavir Treatment Between 95 and 120 Percent at Week 8
Time Frame: week 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 24 | 34 | 21 | 28
participants
  Compliance | 16 | 21 | 13 | 10
  Non-compliance | 8 | 13 | 8 | 18

23. Secondary Outcome: Number Patients With Compliance With Tipranavir Treatment Between 95 and 120 Percent at Week 16
Time Frame: week 16
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 34 | 19 | 26
participants
  Compliance | 16 | 20 | 10 | 13
  Non-compliance | 9 | 14 | 9 | 13

24. Secondary Outcome: Number Patients With Compliance With Tipranavir Treatment Between 95 and 120 Percent at Week 24
Time Frame: week 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 34 | 16 | 25
participants
  Compliance | 17 | 17 | 6 | 14
  Non-compliance | 8 | 17 | 10 | 11

25. Secondary Outcome: Number Patients With Compliance With Tipranavir Treatment Between 95 and 120 Percent at Week 48
Time Frame: week 48
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 24 | 29 | 13 | 22
participants
  Compliance | 19 | 11 | 5 | 11
  Non-compliance | 5 | 18 | 8 | 11

26. Primary Outcome: Number of Severe (DAIDS Grades 3 or 4) Adverse Events Related to Drug for Treated Patients by Age Group and Formulation
Description: Intensity of adverse events were graded by the investigator based on the DAIDS standardized table (Division of AIDS, National Institute of Health). DAIDS Grade 3 (Severe) and Grade 4 (Life Threatening) were identified.
Time Frame: up to 288 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- TPV SEDDS 6-<12 Yrs: Patients treated with Tipranavir SEDDS, ages 6-11
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 6-<12 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 31 | 19 | 6 | 34
participants
  Total with any severe drug-related adverse events | 2 | 6 | 3 | 2 | 5
  Gamma-glutamyl transferase increased | 1 | 2 | 2 | 2 | 1
  Alanine aminotransferase increased | 0 | 1 | 0 | 1 | 4
  Liver function test abnormal | 0 | 1 | 0 | 0 | 0
  Hepatic enzyme abnormal | 0 | 1 | 0 | 0 | 0
  Anemia | 0 | 0 | 1 | 0 | 0
  Nausea | 0 | 1 | 0 | 0 | 0
  Hyperamylasemia | 1 | 0 | 0 | 0 | 0

27. Primary Outcome: Number of Patients With Severe (DAIDS Grades 3 or 4) Laboratory Abnormalities by Age Group and Formulation
Description: as for outcome 26
Time Frame: up to 288 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 6-<12 Yrs | TPV SEDDS 12-18 Yrs
Number analyzed (Participants) | 25 | 30 | 17 | 6 | 34
participants
  Creatinine phosphokinase increased | 4 | 1 | 3 | 0 | 10
  Gamma-glutamyl transferase increased | 4 | 4 | 2 | 2 | 3
  Sodium increased | 2 | 3 | 0 | 4 | 4
  Alanine aminotransferase increased | 0 | 2 | 0 | 3 | 6
  Amylase increased | 2 | 4 | 3 | 0 | 1
  Urine blood | 0 | 0 | 1 | 0 | 4
  Hemoglobin | 0 | 0 | 1 | 0 | 2
  Cholesterol increased | 0 | 0 | 1 | 0 | 2
  Glucose increased | 0 | 0 | 1 | 0 | 2
  Triglyceride increased | 0 | 1 | 1 | 0 | 2
  Calcium decreased | 0 | 2 | 0 | 0 | 0
  Neutrophil count decreased | 0 | 1 | 1 | 0 | 0
  Prothombin time prolonged | 1 | 1 | 0 | 0 | 0
  Partial thromboplastin time prolonged | 1 | 0 | 0 | 0 | 0
  Sodium decreased | 0 | 1 | 0 | 0 | 0
  Potassium increased | 0 | 1 | 0 | 0 | 0
  Potassium decreased | 0 | 0 | 1 | 0 | 0
  Calcium increased | 1 | 0 | 1 | 0 | 2
  Aspartate aminotransferase increased | 0 | 1 | 0 | 0 | 0
  Platelets | 1 | 0 | 0 | 0 | 0
  Urine protein | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Entire study (18Feb2004 to 30Jun2010)
Arm/Group | TPV OS 2-<6 Yrs | TPV OS 6-<12 Yrs | TPV OS 12-18 Yrs | TPV SEDDS 6-<12 Yrs | TPV SEDDS 12-18 Yrs
Serious Adverse Events (participants affected / at risk) | 10/25 | 13/31 | 8/19 | 1/6 | 7/34
Other Adverse Events (participants affected / at risk) | 14/25 | 18/31 | 10/19 | 5/6 | 27/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TPV OS 2-<6 Yrs (N=25) | TPV OS 6-<12 Yrs (N=31) | TPV OS 12-18 Yrs (N=19) | TPV SEDDS 6-<12 Yrs (N=6) | TPV SEDDS 12-18 Yrs (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 2 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Coagulation time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Investigation (Investigations) | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Psychiatric investigation (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Hallucinations, mixed (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophageal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Psychosomatic disease (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TPV OS 2-<6 Yrs (N=25) | TPV OS 6-<12 Yrs (N=31) | TPV OS 12-18 Yrs (N=19) | TPV SEDDS 6-<12 Yrs (N=6) | TPV SEDDS 12-18 Yrs (N=34)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 3 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 5 | 3 | 3 | 0 | 3
Eye pruritus (Eye disorders) | 0 | 2 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 2 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 11 | 2 | 1 | 11
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
Malocclusion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 4 | 1 | 10
Parotid gland enlargement (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 14 | 11 | 5 | 2 | 15
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 2 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 2
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 9 | 8 | 6 | 1 | 9
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Adenovirus infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Body tinea (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 0 | 3
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 6 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 5 | 0 | 0 | 0 | 3
HIV infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Impetigo (Infections and infestations) | 1 | 2 | 1 | 0 | 1
Influenza (Infections and infestations) | 3 | 3 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 6 | 5 | 1 | 0 | 8
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 3 | 3 | 0 | 5
Oral herpes (Infections and infestations) | 2 | 4 | 0 | 0 | 5
Otitis externa (Infections and infestations) | 2 | 3 | 2 | 0 | 0
Otitis media (Infections and infestations) | 6 | 4 | 1 | 1 | 1
Otitis media acute (Infections and infestations) | 4 | 3 | 1 | 0 | 0
Parotitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 5 | 5 | 2 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 1 | 1 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 3 | 1 | 0 | 4
Sinusitis (Infections and infestations) | 9 | 2 | 0 | 1 | 1
Skin candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 5 | 1 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 9 | 7 | 2 | 2 | 6
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 3 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 5 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 6
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 3 | 2 | 4
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 5
Epiphyses delayed fusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 4
Headache (Nervous system disorders) | 2 | 7 | 4 | 1 | 4
Mental impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Mental disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Enuresis (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 13 | 3 | 3 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 4 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1 | 5
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.